CLINICAL TRIAL: NCT05073432
Title: A Study in Development of a Personalized Discussion Prioritization Tool for Older Adults Considering Adjuvant Chemotherapy for Breast Cancer
Brief Title: Development of a Personalized Discussion Prioritization Tool for Older Adults Considering Adjuvant Chemotherapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Allison Magnuson, Assistant Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS20110
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Discussion Prioritization Tool (DPT)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Electronic completion of Geriatric Assessment and Conjoint Analysis with result output.
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — Usability of the Discussion Prioritization Tool (DPT) by completing Geriatric Assessment and Conjoint Analysis

SUMMARY:
The investigators have developed a Discussion Prioritization Tool (DPT) for older adults consider adjuvant chemotherapy that utilizes Conjoint Analysis (CA) methodology and the objective of the current study is to assess usability of this DPT in the target population, older adults with breast cancer and to adapt the tool to optimize usability for the target population.

DETAILED DESCRIPTION:
Given the complexity of adjuvant chemotherapy decision making for older adults with breast cancer, enhancing support and promoting treatment discussions in the context of patient's goals and preferences is an important need. With this need in mind, the investigators have completed interviews with patients with cancer patients who are considering adjuvant therapy. As a result of these interviews, the investigators have developed a common list of attributes (variables found to be important in decision making) that were used to create the Discussion Prioritization Tool (DPT) using Conjoint Analysis (CA) methodology. CA which is a method that can assess the relative importance that patients place on different aspects of care by asking patients to make a series of trade-offs between competing options. The purpose of this study is to assess the usability of a Discussion Prioritization Tool, administered through a tablet, laptop, or computer, for its ability to aid in treatment decision-making. The investigators would like to gather feedback from individuals to improve and adapt the communication tool.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65
* Diagnosis of stage I-III BC
* Being considered for adjuvant chemotherapy
* Able to speak and read English
* Able to participate in study procedures.

Exclusion Criteria:

* Lacking medical decision-making capacity as determined by their oncologist
* Evidence of metastatic disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Magnuson, DO, Principal Investigator — Univ. of Rochester Wilmot Cancer Center
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Functional Assessment of the Discussion Prioritization Tool (DPT)
Description: System Usability Scale (SUS) (score on a 10-item scale, with a total score ranging from 0-100; a higher score corresponds to greater usability). We will deem the tool usable if our mean SUS score among the 10 patients enrolled is >68.
Time Frame: 2 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 10
score on a scale | 78.5 (26.5)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT05073432/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT05073432/ICF_001.pdf